CLINICAL TRIAL: NCT02485639
Title: Analysis of Bone Marrow and Blood B Cell Immune Responses to Influenza Vaccination
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study was terminated due to CoronaVIrus Disease of 2019 (COVID-19) pandemic.
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 14-0059; HHSN272201400004C
Record Dates: First submitted 2015-06-11; First posted 2015-06-30 (Estimated); Results first posted 2023-10-24 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2021-03

CONDITIONS: Influenza; Influenza Immunisation
Keywords: HA (hemagglutinin) -specific plasmablasts; humoral immunity; influenza; memory B cells
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Influenza Virus Vaccine Inactivated (Experimental): All study participants received licensed inactivated influenza vaccine intramuscularly (IM) on Day 0.
  Interventions: Biological: Influenza Virus Vaccine Inactivated

INTERVENTIONS:
Biological: Influenza Virus Vaccine Inactivated — A synthetic vaccine consisting of three inactivated influenza viruses: two different influenza type A strains and one influenza type B strain. Trivalent influenza vaccine is formulated annually, based on influenza strains projected to be prevalent in the upcoming flu season. All participants received vaccine intramuscularly (IM) on Day 0.

SUMMARY:
This was a Phase IV open label and single arm study, with the aim of enrolling up to 55 healthy males and non-pregnant females in a single site, age 18-49 years old, inclusive. This study was designed to assess the humoral response to influenza vaccination and the longevity of humoral immunity to influenza vaccination in healthy adults. Total enrollment was 27 participants.

This was a multi-year study. After one year of participation, participants were offered the opportunity to participate in the study for up to 3 consecutive years, provided eligibility criteria was met each year. Participants who elected to continue in the study after first year of participation were rescreened to verify continued eligibility and re-consented prior to subsequent participation. The primary study objective was to investigate the longevity of humoral immunity to influenza virus in humans.

Note: Due to the Coronavirus Disease of 2019 (COVID-19) pandemic, all non-essential research was halted in mid-March 2020. New enrollments were placed on hold for this study. Follow-up visits were also halted, which impacted the timing of participants' subsequent follow-up visits. Participant visits for Day 7 and Day 14 were not impacted. For this study, there were participants whose Day 28 and Day 90 visits were impacted by the temporary halting of non-essential research studies. As such, a request was submitted to the Emory University Institutional Review Board to extend the missed visit windows for the Day 28 and Day 90 visits for a maximum of up to 180 days, to ensure that ample time was available to bring participants back for their missed visits. Enrollment for this study ended on March 31, 2020, before research activities could resume at Emory.

DETAILED DESCRIPTION:
This was a Phase IV open label and single arm study, with the aim of enrolling up to 55 healthy males and non-pregnant females in a single site, age 18-49 years old, inclusive. This study was designed to assess the humoral response to influenza vaccination and the longevity of humoral immunity to influenza vaccination in healthy adults. Total enrollment was 27 participants.

The laboratory technique used in this study characterized persistence and clonotype of antigen specific B-cells and plasmablasts in blood and bone marrow. Enrolled participants received licensed seasonal inactivated influenza vaccine (administered as a part of the study). The vaccine was administered according to the package insert, and study participants donated serial samples of blood and bone marrow aspirate for immunology monitoring.

Safety was assessed from the time of study enrollment through the last study visit, via monitoring of vital signs, change in health status, and targeted physical exam with safety labs prior to each bone marrow aspirate procedure. Repeated measurements of humoral immunity were obtained at 7 days, 14 days, 28 days, 90 days and at one year post-vaccination to assess the magnitude, clonal diversity and persistence of B-cell responses to influenza vaccination.

This was a multi-year study. After one year of participation, participants were offered the opportunity to participate in the study for up to 3 consecutive years, provided eligibility criteria was met each year. Participants who elected to continue in the study after first year of participation were rescreened to verify continued eligibility and re-consented prior to subsequent participation.

Re-enrolling participants received new subject identifiers and will count towards the total enrollment number for subsequent years of participation. A separate subject record will be maintained each year a subject re-enrolls in the study. Enrollment for the next year will begin with the availability of the seasonal flu vaccine. For participants who elect to re-enroll in the study, the Day 365 visit (+/- 3 month window) would also be the Day 0 visit for the subsequent year. The primary study objective is to investigate the longevity of humoral immunity to influenza virus in humans. The secondary study objective is the longitudinal tracking of vaccine-induced B cell responses with special emphasis on broadly neutralizing HA (hemagglutinin) stem-reactive responses.

Note: Due to the Coronavirus Disease of 2019 (COVID-19) pandemic, all non-essential research was halted in mid-March 2020. New enrollments were placed on hold for this study. Follow-up visits were also halted, which impacted the timing of participants' subsequent follow-up visits. Participant visits for Day 7 and Day 14 were not impacted. For this study, there are participants whose Day 28 and Day 90 visits were impacted by the temporary halting of non-essential research studies. As such, a request was submitted to the Emory University Institutional Review Board to extend the missed visit windows for the Day 28 and Day 90 visits for a maximum of up to 180 days, to ensure that ample time was available to bring participants back for their missed visits. Enrollment for this study ended on March 31, 2020, before research activities could resume at Emory.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant female subjects between 18 and 49 years of age (inclusive).
* Subjects capable of providing written informed consent prior to initiation of any study procedures.
* Subjects able to understand and comply with planned study procedures and be available for all study visits.
* Safety labs:
* White blood cell count (WBC), within reference range of lower limit of normal of 4,000 per microliter (uL), and upper limit of normal of 10,000 per microliter (uL).
* Hemoglobin, within reference range of lower limit of normal of 11.4 grams per deciliter (gm/dL) and upper limit of normal of 16.1 grams per deciliter (gm/dL).
* Hematocrit, within reference range of lower limit of normal of 33.3 percent and an upper limit of normal of 46.5 percent.
* Platelet Count, within reference range of lower limit of normal of 150,000 per microliter (uL) and upper limit of normal of 400,000 per microliter (uL).
* Prothrombin Time (PT/INR), PT below or equal to the upper limit of normal of 13.1 seconds; International Normalized Ratio (INR) within normal reference range of less than 1.5 (normal range for non-anti-coagulated patients).
* Creatinine within reference range of lower limit of normal of 0.4 milligrams per deciliter (mg / dL) and upper limit of normal of 1.2 milligrams per deciliter (mg / dL).
* Potassium, within reference range of lower limit of normal of 3.6 millimolar (mM) and upper limit of normal of 5.1 millimolar (mM).
* Heart rate > / = 55 to < / = 100 per minute.
* Systolic blood pressure > / = 90 to < / = 150 millimeters of mercury (mmHg).
* Diastolic blood pressure < 90 millimeters of mercury (mmHg).
* Oral temperature < 100 degrees Fahrenheit.
* Respirations even, unlabored, and > 10 / minute to < 20 / minute.
* Female subjects of child bearing potential must have a negative urine pregnancy test at the screening visit, enrollment visit and prior to subsequent bone marrow aspirate procedures. Female subjects of childbearing potential must agree to practice abstinence, use a barrier method of birth control, or use an U.S. Food and Drug Administration (FDA) approved form of birth control.
* Subjects who have not received seasonal flu vaccine for the current year (September - June).

Exclusion Criteria:

* If female, active pregnancy or breast-feeding or plans to become pregnant during study participation.
* Subject report of having any medical disease or condition that, in the opinion of the site principal investigator or appropriate sub-investigator, is a contraindication to study participation. This includes any acute or chronic medical disease or condition, defined as persisting 3 months (defined as 90 days) or longer, that would place the subject at an unacceptable risk of injury, render the subject unable to meet the requirements of the protocol, or may interfere with the evaluation of responses or the subject's successful completion of this study.
* Subject report of taking anticoagulants, or long-term (greater than 14 days) systemic steroids or other immunosuppressive medications.
* Subject report of known allergy to lidocaine.
* Subject report of known hypersensitivity or allergy to eggs, egg or chicken protein, report of allergy to components of the study vaccine or other components of the study vaccine.
* Subject report of known latex allergy.
* Subject report of a history of severe reactions following previous immunization with licensed or unlicensed influenza virus vaccines.
* Subject report of a history of Guillain-Barre syndrome.
* Subjects who believe they cannot tolerate the bone marrow aspirations without sedation.
* Subjects with an active infection or that have an acute illness within 72 hours prior to study vaccination. Subject having had an acute illness which is nearly resolved with only minor residual symptoms remaining is allowable if, in the opinion of the site principal investigator or appropriate sub-investigator, the residual symptoms will not interfere with the ability to assess safety parameters as required by the protocol.
* Subjects who are participating in another clinical trial involving the use of investigational agents or vaccines.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2015-12-23 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edmund K Waller, MD, PhD, Principal Investigator — Emory University
Locations (1):
- Emory Clinic - Winship Cancer Institute, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thompson WW, Shay DK, Weintraub E, Brammer L, Cox N, Anderson LJ, Fukuda K. Mortality associated with influenza and respiratory syncytial virus in the United States. JAMA. 2003 Jan 8;289(2):179-86. doi: 10.1001/jama.289.2.179. PMID 12517228
- [Background] Centers for Disease Control and Prevention (CDC). Prevention and control of seasonal influenza with vaccines. Recommendations of the Advisory Committee on Immunization Practices--United States, 2013-2014. MMWR Recomm Rep. 2013 Sep 20;62(RR-07):1-43. PMID 24048214
- [Background] Kunzel W, Glathe H, Engelmann H, Van Hoecke C. Kinetics of humoral antibody response to trivalent inactivated split influenza vaccine in subjects previously vaccinated or vaccinated for the first time. Vaccine. 1996 Aug;14(12):1108-10. doi: 10.1016/0264-410x(96)00061-8. PMID 8911005
- [Background] Pica N, Palese P. Toward a universal influenza virus vaccine: prospects and challenges. Annu Rev Med. 2013;64:189-202. doi: 10.1146/annurev-med-120611-145115. PMID 23327522
- [Background] Wrammert J, Smith K, Miller J, Langley WA, Kokko K, Larsen C, Zheng NY, Mays I, Garman L, Helms C, James J, Air GM, Capra JD, Ahmed R, Wilson PC. Rapid cloning of high-affinity human monoclonal antibodies against influenza virus. Nature. 2008 May 29;453(7195):667-71. doi: 10.1038/nature06890. Epub 2008 Apr 30. PMID 18449194
- [Background] Slifka MK, Antia R, Whitmire JK, Ahmed R. Humoral immunity due to long-lived plasma cells. Immunity. 1998 Mar;8(3):363-72. doi: 10.1016/s1074-7613(00)80541-5. PMID 9529153

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The following methods were used to recruit participants: traditional flyers posted throughout campus, word of mouth referrals, and social media posts. In addition, listserves, and campus newsletters were also leveraged to expand our participant reach.
Groups:
- Influenza Virus Vaccine - Inactivated: All study participants received licensed inactivated influenza vaccine intramuscularly (IM) on Day 0.
  Influenza Virus Vaccine Inactivated: A synthetic vaccine consisting of three inactivated influenza viruses: two different influenza type A strains and one influenza type B strain. Trivalent influenza vaccine is formulated annually, based on influenza strains projected to be prevalent in the upcoming flu season. All participants received vaccine IM on Day 0.
Period: Overall Study
Arm/Group | Influenza Virus Vaccine - Inactivated
Started | 27
Completed | 11
Not Completed | 16
Not completed — 8 participants did not complete study. Study halted due to CoronaVIrus Disease COVID-19 pandemic. | 8
Not completed — Early termination | 4
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Groups:
- Influenza Virus Vaccine - Inactivated: All study participants received licensed inactivated influenza vaccine intramuscularly on Day 0.
  Influenza Virus Vaccine Inactivated: A synthetic vaccine consisting of three inactivated influenza viruses: two different influenza type A strains and one influenza type B strain. Trivalent influenza vaccine is formulated annually, based on influenza strains projected to be prevalent in the upcoming flu season. All participants received vaccine IM on Day 0.
Arm/Group | Influenza Virus Vaccine - Inactivated
Number analyzed (Participants) | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 27
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 27.4 [18 to 49]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 27
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: Number of Influenza-specific Antibody Secreting Cells (ASC) Present in the Blood
Description: Blood Immunoglobulin G (IgG) ASC specific for the seasonal influenza vaccine were measured by enzyme-linked immunosorbent spot (ELISPOT) using vaccine-coated plates. Numbers of influenza-specific ASC per million peripheral blood mononuclear cells are reported.
Time Frame: Day 7
Population: Of the 27 donors enrolled in this study, 24 participants were included in this analysis, as one participant withdrew from the study prior to the Day 7 sample collection, one participant had a failed ELISPOT assay/bad plate batch, and for the remaining donor, a sample was not collected at this time-point, as the donor missed their appointment.
Measure: Geometric Mean (Inter-Quartile Range); unit: Number of Influenza-specific ASC/million
Arm/Group | Influenza Virus Vaccine - Inactivated
Number analyzed (Participants) | 24
Number of Influenza-specific ASC/million | 284.2 [81.8 to 501.2]

2. Primary Outcome: Number of Influenza-specific Antibody Secreting Cells (ASC) Present in the Bone Marrow
Description: Influenza-specific IgG ASC and total IgG ASC were measured in bone marrow samples by ELISPOT using plates coated with influenza vaccine or total IgG capture antibody. Influenza-specific bone marrow IgG ASC numbers are expressed as a percentage of the total bone marrow IgG ASC number.
Time Frame: Day 0
Population: Of the 27 donors enrolled in this study, 15 donors were eligible to have their samples analyzed for this Day 0 time-point outcome measure. 15 participants were analyzed for this time-point outcome measure as due to limited bone marrow yields, as ELISPOT assays were not run on every bone marrow sample. This was the case for 12 of the donors for this time-point outcome measure.
Measure: Geometric Mean (Inter-Quartile Range); unit: Percent of total BM IgG ASC number
Arm/Group | Influenza Virus Vaccine - Inactivated
Number analyzed (Participants) | 15
Percent of total BM IgG ASC number | 1.08 [0.79 to 1.71]

3. Primary Outcome: Number of Influenza-specific Antibody Secreting Cells (ASC) Present in the Bone Marrow
Description: as for outcome 2
Time Frame: Day 28
Population: Of the 27 donors enrolled in this study, 9 donors were eligible to have their samples analyzed for this Day 28 time-point outcome measure. Due to limited bone marrow yields, ELISPOT assays were not run on every bone marrow sample. This was the case for 14 of the donors for this time-point measure. There were two donor/participant withdrawals prior to the Day 28 time-point collection, and two donors were unable to provide a sample, as their lab values were out of range for the bone marrow draw.
Measure: Geometric Mean (Inter-Quartile Range); unit: Percent of total BM IgG ASC number
Arm/Group | Influenza Virus Vaccine - Inactivated
Number analyzed (Participants) | 9
Percent of total BM IgG ASC number | 3.49 [2.19 to 3.75]

4. Primary Outcome: Number of Influenza-specific Antibody Secreting Cells (ASC) Present in the Bone Marrow
Description: as for outcome 2
Time Frame: Day 365
Population: Of the 27 donors enrolled in this study, seven donors were eligible to have their samples analyzed for this Day 365 time-point outcome measure. Due to limited bone marrow yields, ELISPOT assays were not run on every bone marrow sample. This was the case for three of the donors for this time-point outcome measure. There were nine donor/participant withdrawals prior to the Day 365 time-point collection. Eight Day 365 visits were halted due to COVID, and samples could not be collected.
Measure: Geometric Mean (Inter-Quartile Range); unit: Percent of total BM IgG ASC number
Arm/Group | Influenza Virus Vaccine - Inactivated
Number analyzed (Participants) | 7
Percent of total BM IgG ASC number | 1.48 [1.24 to 1.78]

5. Primary Outcome: Number of Influenza-specific Memory B Cells Present in the Blood
Description: Influenza-specific memory B cells were assayed by ELISPOT after polyclonal stimulation of peripheral blood mononuclear cells to generate ASC. The influenza-specific memory B cell frequencies are reported as the percentage of IgG secreting cells found in the stimulated cultures.
Time Frame: Day 0
Population: Of the 27 donors enrolled in this study, all 27 donors were eligible to have their samples analyzed for this Day 0 time-point outcome measure.
Measure: Geometric Mean (Inter-Quartile Range); unit: percentage of IgG secreting cells
Arm/Group | Influenza Virus Vaccine - Inactivated
Number analyzed (Participants) | 27
percentage of IgG secreting cells | .81 [.60 to 1.34]

6. Primary Outcome: Number of Influenza-specific Memory B Cells Present in the Blood
Description: as for outcome 5
Time Frame: Day 28
Population: Of the 27 donors enrolled in this study, 25 donors were eligible to have their samples analyzed for this Day 28 time-point outcome measure. There were two donor withdrawals prior to the Day 28 time-point collection.
Measure: Geometric Mean (Inter-Quartile Range); unit: percentage of IgG secreting cells
Arm/Group | Influenza Virus Vaccine - Inactivated
Number analyzed (Participants) | 25
percentage of IgG secreting cells | 2.3 [1.35 to 4.40]

7. Primary Outcome: Number of Influenza-specific Memory B Cells Present in the Blood
Description: as for outcome 5
Time Frame: Day 365
Population: Of the 27 donors enrolled in this study, 10 donors were eligible to have their samples analyzed for this Day 365 time-point outcome measure. There were 9 donor/participant withdrawals prior to the Day 365 time-point collection. COVID halted the Day 365 visits for 8 participants.
Measure: Geometric Mean (Inter-Quartile Range); unit: percentage of IgG secreting cells
Arm/Group | Influenza Virus Vaccine - Inactivated
Number analyzed (Participants) | 10
percentage of IgG secreting cells | 0.82 [0.49 to 1.49]

8. Primary Outcome: Number of Subjects Who Initially Seroconverted and Maintained Seroconversion at 1 Year Post Vaccination
Description: Initial seroconversion is defined as having a pre-vaccination (day 0) hemagglutination inhibition (HAI) titer < 1:40 against a particular strain and a day 28 post-vaccination titer > / = 1:40 against the same strain OR a pre-vaccination HAI titer >1:40 and an increase in titer of at least 4-fold on day 28 relative to day 0. Maintenance of seroconversion in those who initially seroconverted is defined as maintaining an HAI titer >/= 40 at 1 year in those with day 0 titers < 40 OR maintaining a >/= 4-fold increase in HAI titer at one year compared to day 0.
  HAI assays were performed using 0.75% guinea pig red blood cells and virus stocks matched to the strains in the vaccines received by each donor.
Time Frame: Day 365
Population: Many of the participants enrolled in the last season of the study were lost to follow-up for the one year timepoint due to research being halted due to COVID.
Measure: Count of Participants; unit: Participants
Arm/Group | Influenza Virus Vaccine - Inactivated
Number analyzed (Participants) | 10
Participants
  H1N1 seroconversion maintenance: never seroconverted | 9
  H1N1 seroconversion maintenance: seroconverted at day 28 but seroconversion not maintained at day 365 | 1
  H1N1 seroconversion maintenance: seroconverted at day 28 and maintained seroconversion at day 365 | 0
  H3N2 seroconversion maintenance: never seroconverted | 9
  H3N2 seroconversion maintenance: seroconverted at day 28 but seroconversion not maintained at day 365 | 0
  H3N2 seroconversion maintenance: seroconverted at day 28 and maintained seroconversion at day 365 | 1
  B/Victoria seroconversion maintenance: never seroconverted | 10
  B/Victoria seroconversion maintenance: seroconverted at day 28 but seroconversion not maintained at day 365 | 0
  B/Victoria seroconversion maintenance: seroconverted at day 28 and maintained seroconversion at day 365 | 0
  B/Yamagata seroconversion maintenance: never seroconverted | 9
  B/Yamagata seroconversion maintenance: seroconverted at day 28 but seroconversion not maintained at day 365 | 0
  B/Yamagata seroconversion maintenance: seroconverted at day 28 and maintained seroconversion at day 365 | 1

9. Primary Outcome: Number of Subjects Achieving Seroconversion to Each of the Strains in the Vaccine
Description: Seroconversion defined as having a pre-vaccination (day 0) hemagglutination inhibition (HAI) titer < 1:40 against a particular strain and a Day 28 post-vaccination titer > / = 1:40 against the same strain OR a pre-vaccination HAI titer >1:40 and an increase in titer of at least 4-fold on day 28. HAI assays were performed using 0.75% guinea pig red blood cells and virus stocks matched to the strains in the vaccines received by each donor.
Time Frame: Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Influenza Virus Vaccine - Inactivated
Number analyzed (Participants) | 25
Participants
  H1N1 seroconversion: HAI < 1:40 on day 0, HAI < 1:40 on day 28 (no seroconversion) | 0
  H1N1 seroconversion: HAI < 1:40 on day 0, HAI >/= 1:40 on day 28 (seroconverted) | 1
  H1N1 seroconversion: HAI >/= 1:40 on day 0, < 4-fold HAI increase on day 28 (no seroconversion) | 20
  H1N1 seroconversion: HAI >/= 1:40 on day 0, >/= 4-fold HAI increase on day 28 (seroconverted) | 4
  H3N2 seroconversion: HAI < 1:40 on day 0, HAI < 1:40 on day 28 (no seroconversion) | 0
  H3N2 seroconversion: HAI < 1:40 on day 0, HAI >/= 1:40 on day 28 (seroconverted) | 5
  H3N2 seroconversion: HAI >/= 1:40 on day 0, < 4-fold HAI increase on day 28 (no seroconversion) | 15
  H3N2 seroconversion: HAI >/= 1:40 on day 0, >/= 4-fold HAI increase on day 28 (seroconverted) | 5
  B/Victoria seroconversion: HAI < 1:40 on day 0, HAI < 1:40 on day 28 (no seroconversion) | 7
  B/Victoria seroconversion: HAI < 1:40 on day 0, HAI >/= 1:40 on day 28 (seroconverted) | 4
  B/Victoria seroconversion: HAI >/= 1:40 on day 0, < 4-fold HAI increase on day 28 (no seroconversion) | 14
  B/Victoria seroconversion: HAI >/= 1:40 on day 0, >/= 4-fold HAI increase on day 28 (seroconverted) | 0
  B/Yamagata seroconversion: HAI < 1:40 on day 0, HAI < 1:40 on day 28 (no seroconversion) | 0
  B/Yamagata seroconversion: HAI < 1:40 on day 0, HAI >/= 1:40 on day 28 (seroconverted) | 1
  B/Yamagata seroconversion: HAI >/= 1:40 on day 0, < 4-fold HAI increase on day 28 (no seroconversion) | 21
  B/Yamagata seroconversion: HAI >/= 1:40 on day 0, >/= 4-fold HAI increase on day 28 (seroconverted) | 3

10. Secondary Outcome: Frequency of Hemagglutinin Stem Reactive Responses to Influenza Vaccine Among Blood Plasmablasts
Description: Blood IgG ASC specific for the seasonal influenza vaccine were measured by ELISPOT using plates coated with chimeric hemagglutinin antigen containing the pandemic H1 stem domain fused to the head domain of an H9 influenza virus. Numbers of stem-specific ASC per million peripheral blood mononuclear cells are reported.
Time Frame: Day 7
Population: Of the 27 donors enrolled in this study, 19 donors were eligible to have their samples analyzed for this Day 7 time-point outcome measure. There was 1 donor/participant withdrawal prior to the Day 7 time-point collection. Three samples were not able to be used due to a failed assay, a processing error and a missed appointment. Due to limited yields, assays were not performed on four of the samples.
Measure: Geometric Mean (Inter-Quartile Range); unit: Number of stem-specific ASC per mil PBMC
Arm/Group | Influenza Virus Vaccine - Inactivated
Number analyzed (Participants) | 19
Number of stem-specific ASC per mil PBMC | 1.24 [.70 to 2.76]

11. Secondary Outcome: Frequency of Hemagglutinin Stem Reactive Responses to Influenza Vaccine Among the Bone Marrow Plasma Cells
Description: Influenza-specific IgG ASC and total IgG ASC were measured in bone marrow samples by ELISPOT using plates coated with H9 head/H1 stem chimeric hemagglutinin antigen or total IgG capture antibody. Stem-specific bone marrow IgG ASC numbers are expressed as a percentage of the total bone marrow IgG ASC number.
Time Frame: Day 365
Population: This assay was not run due to limited sample quantities.
Arm/Group | Influenza Virus Vaccine - Inactivated
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 year Adverse event data were collected from Day 0 (enrollment) to Day 365 (the end of follow-up). Adverse event data were collected at each of the follow-up visits (Day 7, Day 14, Day 28, Day 90, and Day 365).
Description: At each of the follow-up visits (Day 7, Day 14, Day 28, Day 90, and Day 365), participants were asked about any adverse events that they might have experienced since their last visit. Clinical health assessments were conducted at every study visit, and included inquiry regarding any illness, any change in medication, and any overall health changes since the last study visit. Adverse event data was collected from enrollment until the end of follow-up at Day 365.
Groups:
- Influenza Virus Vaccine Inactivated: All study participants received licensed inactivated influenza vaccine intramuscularly on Day 0.
  Influenza Virus Vaccine Inactivated: A synthetic vaccine consisting of three inactivated influenza viruses: two different influenza type A strains and one influenza type B strain. Trivalent influenza vaccine is formulated annually, based on influenza strains projected to be prevalent in the upcoming flu season. All participants received vaccine IM on Day 0.
Arm/Group | Influenza Virus Vaccine Inactivated
All-Cause Mortality (participants affected / at risk) | 0/27
Serious Adverse Events (participants affected / at risk) | 0/27
Other Adverse Events (participants affected / at risk) | 1/27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Influenza Virus Vaccine Inactivated (N=27)
Nausea (Gastrointestinal disorders) | 1 (1) — Mild nausea reported by participant. Onset and end date of mild nausea was 2/17/2016. Deemed not related to study. Participant recovered completely. Not a Serious Adverse Event. No action taken.

LIMITATIONS AND CAVEATS:
Due to the COVID-19 pandemic, all non-essential research was halted at our site (mid-March 2020). New enrollments and follow-up visits were halted, impacting participants' follow-up visits. One Day 28 visit was halted, three Day 90 visits were halted. Seven Day 365 visits were halted. We requested an expansion of the visit windows, however, enrollment for this study ended on March 31, 2020, before research activities could resume at Emory.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-06-04): https://cdn.clinicaltrials.gov/large-docs/39/NCT02485639/Prot_SAP_000.pdf
  • Informed Consent Form (2021-01-21): https://cdn.clinicaltrials.gov/large-docs/39/NCT02485639/ICF_001.pdf